CLINICAL TRIAL: NCT00763516
Title: A Pilot Study Using Neoadjuvant Proton Beam Radiation Therapy and Chemotherapy for Marginally Resectable Carcinoma of the Pancreas
Brief Title: Proton Radiation for Resectable Carcinoma of the Pancreas
Acronym: PC02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0704-PC02
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Proton radiation; Chemotherapy; Xeloda; Gemzar; Resectable; Surgery
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiation and chemotherapy (Experimental): Proton radiation
  Capecitabine chemotherapy on radiation days
  Surgery
  Gemcitabine chemotherapy
  Interventions: Radiation: Proton radiation and chemotherapy

INTERVENTIONS:
Radiation: Proton radiation and chemotherapy — Neoadjuvant Chemotherapy Capecitabine (Xeloda®) 1,000 mg by mouth twice a day 5 days/week (M-F) on radiation days only
  Proton radiation 50.4 cobalt gray equivalent(CGE) in 28 fractions over 6 weeks
  Surgery: Gross total resection of primary tumor and regional lymph nodes done 6 weeks after completion of radiation
  Adjuvant Chemotherapy starting 2-8 weeks after surgery Suggested Regimen: Gemcitabine (Gemzar®) 1,000 mg/m2 IV total of 18 doses
  Other Names: Xeloda; Gemzar

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, proton radiation combined with chemotherapy and surgery has on you and your pancreatic cancer. This study will look at the side effects from the treatment and the quality of your life in relation to pain. It will also look at how the tumor responds to the combination of treatment with radiation, chemotherapy and surgery.

DETAILED DESCRIPTION:
Chemotherapy capecitabine on radiation days

Proton radiation over 6 weeks

Surgery 6 weeks after radiation completion

Adjuvant Chemotherapy starting 2-8 weeks after surgery with Gemzar

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas.
* Patients must have marginally resectable disease.
* Patients with biliary obstruction must have adequate drainage prior to starting chemoradiation.

Exclusion Criteria:

* Evidence of distant metastasis including peritoneal seeding and/or ascites.
* Previous irradiation to the abdomen that would compromise the ability to deliver the prescribed treatment.
* Prior surgical resection.
* Gastroduodenal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of grade 3+ bowel perforation, grade 3+ bleeding and grade 4+ nonhematologic acute adverse events (occuring within 90 days of treatment start) | 1 year following the completion of radiation therapy

SECONDARY OUTCOMES:
Collect and analyze tumor control outcomes | 1 year following the completion of radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Romaine C Nichols, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saif MW. Pancreatic cancer: highlights from the 42nd annual meeting of the American Society of Clinical Oncology, 2006. JOP. 2006 Jul 10;7(4):337-48. PMID 16832131
- [Background] Bramhall SR, Allum WH, Jones AG, Allwood A, Cummins C, Neoptolemos JP. Treatment and survival in 13,560 patients with pancreatic cancer, and incidence of the disease, in the West Midlands: an epidemiological study. Br J Surg. 1995 Jan;82(1):111-5. doi: 10.1002/bjs.1800820137. PMID 7881926
- [Background] Klinkenbijl JH, Jeekel J, Sahmoud T, van Pel R, Couvreur ML, Veenhof CH, Arnaud JP, Gonzalez DG, de Wit LT, Hennipman A, Wils J. Adjuvant radiotherapy and 5-fluorouracil after curative resection of cancer of the pancreas and periampullary region: phase III trial of the EORTC gastrointestinal tract cancer cooperative group. Ann Surg. 1999 Dec;230(6):776-82; discussion 782-4. doi: 10.1097/00000658-199912000-00006. PMID 10615932
- [Background] Further evidence of effective adjuvant combined radiation and chemotherapy following curative resection of pancreatic cancer. Gastrointestinal Tumor Study Group. Cancer. 1987 Jun 15;59(12):2006-10. doi: 10.1002/1097-0142(19870615)59:123.0.co;2-b. PMID 3567862
- [Background] Neoptolemos JP, Stocken DD, Friess H, Bassi C, Dunn JA, Hickey H, Beger H, Fernandez-Cruz L, Dervenis C, Lacaine F, Falconi M, Pederzoli P, Pap A, Spooner D, Kerr DJ, Buchler MW; European Study Group for Pancreatic Cancer. A randomized trial of chemoradiotherapy and chemotherapy after resection of pancreatic cancer. N Engl J Med. 2004 Mar 18;350(12):1200-10. doi: 10.1056/NEJMoa032295. PMID 15028824
- [Background] Spitz FR, Abbruzzese JL, Lee JE, Pisters PW, Lowy AM, Fenoglio CJ, Cleary KR, Janjan NA, Goswitz MS, Rich TA, Evans DB. Preoperative and postoperative chemoradiation strategies in patients treated with pancreaticoduodenectomy for adenocarcinoma of the pancreas. J Clin Oncol. 1997 Mar;15(3):928-37. doi: 10.1200/JCO.1997.15.3.928. PMID 9060530
- [Background] Neoptolemos JP, Stocken DD, Dunn JA, Almond J, Beger HG, Pederzoli P, Bassi C, Dervenis C, Fernandez-Cruz L, Lacaine F, Buckels J, Deakin M, Adab FA, Sutton R, Imrie C, Ihse I, Tihanyi T, Olah A, Pedrazzoli S, Spooner D, Kerr DJ, Friess H, Buchler MW; European Study Group for Pancreatic Cancer. Influence of resection margins on survival for patients with pancreatic cancer treated by adjuvant chemoradiation and/or chemotherapy in the ESPAC-1 randomized controlled trial. Ann Surg. 2001 Dec;234(6):758-68. doi: 10.1097/00000658-200112000-00007. PMID 11729382
- [Background] Sohn TA, Yeo CJ, Cameron JL, Koniaris L, Kaushal S, Abrams RA, Sauter PK, Coleman J, Hruban RH, Lillemoe KD. Resected adenocarcinoma of the pancreas-616 patients: results, outcomes, and prognostic indicators. J Gastrointest Surg. 2000 Nov-Dec;4(6):567-79. doi: 10.1016/s1091-255x(00)80105-5. PMID 11307091
- [Background] Brunner TB, Grabenbauer GG, Meyer T, Golcher H, Sauer R, Hohenberger W. Primary resection versus neoadjuvant chemoradiation followed by resection for locally resectable or potentially resectable pancreatic carcinoma without distant metastasis. A multi-centre prospectively randomised phase II-study of the Interdisciplinary Working Group Gastrointestinal Tumours (AIO, ARO, and CAO). BMC Cancer. 2007 Mar 6;7:41. doi: 10.1186/1471-2407-7-41. PMID 17338829
- [Background] Yoshida T, Matsumoto T, Sasaki A, Shibata K, Aramaki M, Kitano S. Outcome of paraaortic node-positive pancreatic head and bile duct adenocarcinoma. Am J Surg. 2004 Jun;187(6):736-40. doi: 10.1016/j.amjsurg.2003.07.031. PMID 15191867
- [Background] Sasson AR, Wetherington RW, Hoffman JP, Ross EA, Cooper H, Meropol NJ, Freedman G, Pingpank JF, Eisenberg BL. Neoadjuvant chemoradiotherapy for adenocarcinoma of the pancreas: analysis of histopathology and outcome. Int J Gastrointest Cancer. 2003;34(2-3):121-8. doi: 10.1385/IJGC:34:2-3:121. PMID 15361645
- [Background] Pingpank JF, Hoffman JP, Ross EA, Cooper HS, Meropol NJ, Freedman G, Pinover WH, LeVoyer TE, Sasson AR, Eisenberg BL. Effect of preoperative chemoradiotherapy on surgical margin status of resected adenocarcinoma of the head of the pancreas. J Gastrointest Surg. 2001 Mar-Apr;5(2):121-30. doi: 10.1016/s1091-255x(01)80023-8. PMID 11331473
- [Background] White RR, Xie HB, Gottfried MR, Czito BG, Hurwitz HI, Morse MA, Blobe GC, Paulson EK, Baillie J, Branch MS, Jowell PS, Clary BM, Pappas TN, Tyler DS. Significance of histological response to preoperative chemoradiotherapy for pancreatic cancer. Ann Surg Oncol. 2005 Mar;12(3):214-21. doi: 10.1245/ASO.2005.03.105. Epub 2005 Mar 3. PMID 15827813
- [Background] Breslin TM, Hess KR, Harbison DB, Jean ME, Cleary KR, Dackiw AP, Wolff RA, Abbruzzese JL, Janjan NA, Crane CH, Vauthey JN, Lee JE, Pisters PW, Evans DB. Neoadjuvant chemoradiotherapy for adenocarcinoma of the pancreas: treatment variables and survival duration. Ann Surg Oncol. 2001 Mar;8(2):123-32. doi: 10.1007/s10434-001-0123-4. PMID 11258776
- [Background] Mackean M, Planting A, Twelves C, Schellens J, Allman D, Osterwalder B, Reigner B, Griffin T, Kaye S, Verweij J. Phase I and pharmacologic study of intermittent twice-daily oral therapy with capecitabine in patients with advanced and/or metastatic cancer. J Clin Oncol. 1998 Sep;16(9):2977-85. doi: 10.1200/JCO.1998.16.9.2977. PMID 9738566
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Bussels B, Goethals L, Feron M, Bielen D, Dymarkowski S, Suetens P, Haustermans K. Respiration-induced movement of the upper abdominal organs: a pitfall for the three-dimensional conformal radiation treatment of pancreatic cancer. Radiother Oncol. 2003 Jul;68(1):69-74. doi: 10.1016/s0167-8140(03)00133-6. PMID 12885454
- [Background] Eccles C, Brock KK, Bissonnette JP, Hawkins M, Dawson LA. Reproducibility of liver position using active breathing coordinator for liver cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):751-9. doi: 10.1016/j.ijrobp.2005.05.066. PMID 16458774
- [Background] Korreman SS, Pedersen AN, Nottrup TJ, Specht L, Nystrom H. Breathing adapted radiotherapy for breast cancer: comparison of free breathing gating with the breath-hold technique. Radiother Oncol. 2005 Sep;76(3):311-8. doi: 10.1016/j.radonc.2005.07.009. PMID 16153728
- [Background] Sugahara S, Tokuuye K, Okumura T, Nakahara A, Saida Y, Kagei K, Ohara K, Hata M, Igaki H, Akine Y. Clinical results of proton beam therapy for cancer of the esophagus. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):76-84. doi: 10.1016/j.ijrobp.2004.04.003. PMID 15629597
- [Background] Gierga DP, Chen GT, Kung JH, Betke M, Lombardi J, Willett CG. Quantification of respiration-induced abdominal tumor motion and its impact on IMRT dose distributions. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1584-95. doi: 10.1016/j.ijrobp.2003.09.077. PMID 15050340
- [Background] Wong JW, Sharpe MB, Jaffray DA, Kini VR, Robertson JM, Stromberg JS, Martinez AA. The use of active breathing control (ABC) to reduce margin for breathing motion. Int J Radiat Oncol Biol Phys. 1999 Jul 1;44(4):911-9. doi: 10.1016/s0360-3016(99)00056-5. PMID 10386650
- [Background] Singh AK, Tierney RM, Low DA, Parikh PJ, Myerson RJ, Deasy JO, Wu CS, Pereira GC, Wahab SH, Mutic S, Grigsby PW, Hope AJ. A prospective study of differences in duodenum compared to remaining small bowel motion between radiation treatments: implications for radiation dose escalation in carcinoma of the pancreas. Radiat Oncol. 2006 Sep 4;1:33. doi: 10.1186/1748-717X-1-33. PMID 16952315
- [Background] Blackall JM, Ahmad S, Miquel ME, McClelland JR, Landau DB, Hawkes DJ. MRI-based measurements of respiratory motion variability and assessment of imaging strategies for radiotherapy planning. Phys Med Biol. 2006 Sep 7;51(17):4147-69. doi: 10.1088/0031-9155/51/17/003. Epub 2006 Aug 8. PMID 16912374
- [Background] Fishman B, Pasternak S, Wallenstein SL, Houde RW, Holland JC, Foley KM. The Memorial Pain Assessment Card. A valid instrument for the evaluation of cancer pain. Cancer. 1987 Sep 1;60(5):1151-8. doi: 10.1002/1097-0142(19870901)60:53.0.co;2-g. PMID 3300951
- [Background] Varadhachary GR, Tamm EP, Abbruzzese JL, Xiong HQ, Crane CH, Wang H, Lee JE, Pisters PW, Evans DB, Wolff RA. Borderline resectable pancreatic cancer: definitions, management, and role of preoperative therapy. Ann Surg Oncol. 2006 Aug;13(8):1035-46. doi: 10.1245/ASO.2006.08.011. Epub 2006 Jul 24. PMID 16865597
- [Background] Ben-Josef E, Shields AF, Vaishampayan U, Vaitkevicius V, El-Rayes BF, McDermott P, Burmeister J, Bossenberger T, Philip PA. Intensity-modulated radiotherapy (IMRT) and concurrent capecitabine for pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):454-9. doi: 10.1016/j.ijrobp.2003.11.019. PMID 15145162
- [Background] Hsiung-Stripp DC, McDonough J, Masters HM, Levin WP, Hahn SM, Jones HA, Metz JM. Comparative treatment planning between proton and X-ray therapy in pancreatic cancer. Med Dosim. 2001 Fall;26(3):255-9. doi: 10.1016/s0958-3947(01)00072-3. PMID 11704461
- [Background] Crane unpublished data presented at ASCO GI, 2006-Abstract # 106; Das, P., et al.).